CLINICAL TRIAL: NCT02620072
Title: Mechanistic Study Using Oral Insulin for Immune Efficacy in Secondary Prevention of Type 1 Diabetes
Brief Title: Fr1da Insulin Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Technische Universität Dresden (Other); Ludwig-Maximilians - University of Munich (Other); Helmholtz Zentrum München (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 808040019
Record Dates: First submitted 2015-11-29; First posted 2015-12-02 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Stage 1 Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; T1D; diabetes mellitus; oral insulin; oral tolerance; autoantigen; self tolerance; prevention; at risk for developing type 1 diabetes; juvenile diabetes; dysglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral insulin capsule (dose escalation using 2 dose strengths) (Experimental): Dose 1 is 7.5 mg rH-insulin crystals; dose 2 is 67.5 mg rH-insulin crystals. Insulin crystals are formulated together with filling substance (microcrystalline cellulose to a total weight of 200 mg) contained in hard gelatine capsules given orally.
  Interventions: Drug: Oral Insulin
- Placebo capsule (Placebo Comparator): Daily administration of placebo capsules containing filling substance (microcrystalline cellulose).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Insulin — Total of 12 months treatment; dose escalation scheme: daily treatment with 7.5 mg or placebo for 3 months; increasing to daily treatment with 67.5 mg or placebo for the following 9 months of the treatment period. Follow-up will continue for 24 months after the last administration of treatment.
  Arms: oral insulin capsule (dose escalation using 2 dose strengths)
Other: Placebo — Total of 12 months intervention period; daily administration of insulin or placebo capsules containing filling substance (microcrystalline cellulose). Follow-up will continue for 24 months after the last administration of treatment.
  Arms: Placebo capsule

SUMMARY:
Type 1 diabetes (T1D) results from an autoimmune destruction of the insulin-producing beta cells. The process of autoimmune destruction is identified by circulating islet autoantibodies to beta cell antigens, and is mediated by a lack of immunological self-tolerance. Self-tolerance is achieved by T cell exposure to antigen in the thymus or periphery in a manner that deletes autoreactive effector T cells or induces regulatory T cells. Immunological tolerance can be achieved by administration of antigen under appropriate conditions. Evidence is now emerging in humans that these approaches may be effective in chronic inflammatory diseases such as multiple sclerosis and allergy. Administration of oral insulin in multiple islet autoantibody-positive children offers the potential for inducing immunological tolerance to beta cells and thereby protect against further development progression to type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is a disease that predominantly affects children. T1D is preceded by islet autoimmunity, which often starts in early childhood and which has a peak incidence at around 1 to 2 years of age. Previous studies show that multiple islet autoantibodies indicate a point of limited return in the path to T1D. Every year, around 10% of multiple islet autoantibody positive children progress from islet autoantibody positivity to symptomatic T1D. Thus, therapy and intervention is needed to change the inevitable path to insulin dependence. Treated should be initiated early when most beta cells are still intact and when the autoimmune process is less advanced may be more effective.

Administration of oral insulin in multiple islet autoantibody-positive children offers the potential for immunological tolerance against beta cells and thereby protect against progression to T1D. Previous studies in rodents had indicated that mucosal administration of insulin is effective in inducing regulatory immune responses that can prevent autoimmune diabetes. Mouse studies indicated that the dose of oral insulin is important. In human studies oral insulin administration shows an excellent safety profile, without adverse side effects at doses between 2.5 and 7.5 mg per day (1-3). The administration of oral insulin (7.5 mg per day) to prediabetic ICA and IAA positive first degree relatives of T1D patients within the DPT-1 study showed no significant beneficial effect in the intention to treat analysis. A sub-analysis of the data, however, showed significant benefit in those relatives with higher titer IAA.

The Pre-POINT study, the first primary autoantigen vaccination dose-finding study in which children with high genetic risk for type 1 diabetes were administered insulin orally daily tested doses (2.5 mg; 7.5 mg; 22.5 mg and 67.5 mg) showed five of six children exposed to a dose of 67.5 mg insulin had evidence of an antibody or T cell response to insulin. The response differed to the typical responses seen in children who develop diabetes in that the antibody responses were of weak affinity and the T cell responses had a preponderance of cells with regulatory T cell phenotypes (37). These results are also encouraging from a safety viewpoint and indicate that oral exposure to insulin at doses that are approximately equivalent to efficacious doses in rodents may promote tolerance in children.

A secondary prevention study using 7.5 mg oral insulin administered daily is currently conducted by the TrialNet Study Group, and includes the Forschergruppe Diabetes, Klinikum rechts der Isar der Technischen Universität München as a study site. Autoantibody, normoglycemic subjects aged 3 to 45 years are treated with oral insulin. In this currently conducted trial there have been no safety issues reported thus far.

The active substance for oral application is human insulin, synthesized in a special non-disease-producing laboratory strain of Escherichia coli bacteria that has been genetically altered by the addition of the gene for human insulin production (Lilly Pharmaceuticals, Indianapolis, Indiana, USA). The physical, chemical and pharmaceutical properties of the human insulin have been well documented by the manufacturer. Oral Insulin will be applied as a capsule containing 7.5 mg of the active substance together with filling substance cellulose and a dose escalation to 67.5 mg of the active substance together with filling substance cellulose. After ingestion, most of the insulin will be degraded by gastric acids. Enteric delivery and systemic availability is therefore unlikely and efficacy of active insulin is likely to be restricted to the oral mucosa.

The Fr1da Insulin Intervention Study intends doses for oral application at 7.5 mg and 67.5 mg per day. The aim of the study is to determine whether daily administration of up to 67.5 mg insulin to young children aged 2 years to 12 years with multiple islet autoantibodies alters the immune responses to insulin over an intervention period of 12 months and whether an altered immune response is associated with protection from developing dysglycemia or diabetes and whether oral insulin treatment reduces the rate of progression to dysglycemia or diabetes.

The immune response to oral insulin treatment has not yet been demonstrated to indicate protection from disease. To address this, the Fr1da Insulin Intervention Study included dysglycemia as a co-primary outcome in the trial, through novel data indicating that dysglycemia is a valid outcome on the path to type 1 diabetes. Once such dysglycemia is present in multiple autoantibody positive subjects, there is an average time of 2 years to clinical symptomatic diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed by either parent(s) or legal guardian(s).
2. Children aged 2 years to 12 years.
3. Positive for at least two islet autoantibodies out of autoantibodies to glutamic acid decarboxylase (GAD65), to insulin (IAA), autoantibodies to IA-2 (IA2A), or autoantibodies to zink transporter 8 (ZnT8A) (time between screening sample collection and randomization must not exceed 90 days).
4. Normoglycemia assessed by oral glucose tolerance test (OGTT).
5. Participation in an observational study that regularly monitors diabetes development

Exclusion Criteria:

Participants meeting any of the following criteria will NOT be eligible for inclusion into the study:

1. dysglycaemia or overt hyperglycemia (diabetes)
2. Concomitant disease or treatment that may interfere with assessment or cause immunosuppression, as judged by the investigators.
3. Current participation in another intervention trial.
4. Any condition that could be associated with poor compliance.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Immune response to insulin | change from baseline (visit 1) to 12 months of treatment
  Immune response measures will be salivary IgA antibodies to insulin, blood CD4+ T cell responses to insulin, and autoantibodies to insulin. Participants are categorized as immune responders if they show a change in at least one of these measures from baseline to 12 months. The number and frequency of immune responders will be compared between the placebo and study drug treatedchildren. If a treatment effect on responder status is observed in the first 90 participants (two-tailed p value <0.05), the responder status will be measured for the remaining participants and the progression to dysglycemia or diabetes will be compared between immune responders and non-responders using Cox proportional hazards model.
Dysglycemia or diabetes | every 6 months up to at least 24 months after baseline
  Dysglycemia is determined through Oral Glucose Tolerance Test (OGTT):
  Dysglycemia is defined as:
  1. Fasting plasma glucose ≥ 110 mg/dL (6.1 mmol/L) and < 126 mg/dL (7 mmol/L), or
  2. 2 hour plasma glucose ≥ 140 mg/dL (7.8 mmol/L) and < 200 (11.1 mmol/L), or
  3. 30, 60, 90 minute plasma glucose during OGTT ≥ 200 mg/dL (11.1 mmol/L)
  Diabetes is defined as:
  1. random blood glucose value ≥200 mg/dl (11.1 mmol/L), or
  2. fasting blood glucose value ≥126 mg/dl (7 mmol/L), or
  3. a 2-hour plasma glucose ≥200 mg/dl (11.1 mmol/L) measured by Oral Glucose Tolerance Test Cox proportional hazards model will be used to compare development of dysglycemia or diabetes between the placebo and study drug treated children.
  For each primary outcome, analyses will also be performed separately in children with the susceptible INS genotype and children with the HLA DR4 allele.

SECONDARY OUTCOMES:
Gene expression of single cells. | Gene expression profile measurement on insulin-responsive cells at 12 month visit
  The FOXP3 signature/IFNG signature ratio of the insulin responsive T-cells will be compared between the placebo and study drug treated children. In addition the expression for a panel of genes in insulin-responsive T cells will be compared between the placebo and study drug treated children.
The change from baseline in insulin autoantibodies | change from baseline to 3 months, 6, months, and 12 months
  The change in insulin autoantibodies will be measured by radio-binding assay. It will be compared between placebo and study drug treated children at the 3 months, 6 months, and 12 months time points using ANOVA and normalized data.
Number of circulating Insulin-tetramer positive T cells | comparison at 9 month visit
  The number of circulating Insulin-tetramer positive CD4+CD25+FOXP3+ T cells (measured at 9 months) will be compared between placebo and study drug treated children using ANOVA.
CD4+ T cell responses to insulin | comparison at 0, 3, 6, and 12 month visit
  The CD4+ T cell response is measured by proliferation assay and will be compared between the placebo and study drug treated children at baseline, 3, 6, and 12 months.
CD8+ T cell responses to insulin | comparison at 0, 3, 6, and 12 month visit
  The CD8+ T cell response is measured by proliferation assay and will be compared between the placebo and study drug treated children at baseline, 3, 6, and 12 months.
Microbiome alpha diversity, beta diversity and taxanomic abundance | comparison at 0, 6, and 12 month visits
  The alpha diversity, beta diversity and taxanomic abundance is measured in stool samples using 16S and metagenomic methods and will be compared between the placebo and study drug treated children at baseline, 6, and 12 months.
Monocyte and T cell sub-populations | comparison at 0, 3, 6, 9, and 12 month visits
  Flow cytometry performed on peripheral blood mononuclear cells to identify monocyte and T cell subpopulations and activated cells based on surface and intracellular markers. The populations will be compared between the placebo and study drug treated children at baseline, 3, 6, 9, and 12 months visits
Plasma inflammatory proteins | comparison at 0, and 12 month visits
  A panel of inflammation proteins measured in plasma by OLINK technology. The quantitative values will be compared between the placebo and study drug treated children at baseline and 12 months.
Transcriptome of peripheral blood mononuclear cells | comparison at 0, and 12 month visits
  The transcriptome of isolated peripheral blood mononuclear cells is measured by RNA seq at baseline and at the 12 month visit. Differentially expressed genes (DEG) and pathway analysis of DEG will be compared between the placebo and study drug treated children at baseline, and 12 months, and between baseline and 12 month visits in study drug and placebo treated children.
Progression to diabetes | Measured at baseline (visit 1) and at each subsequent visit of the treatment phase (visits 2, 3, 4, 5) and observational follow-up of 24 to 54 months after the one year treatment (visits 6, 7, 8, 9, 10, 11, 12, 13, 14)
  Diabetes is defined as:
  1. random blood glucose value ≥200 mg/dl (11.1 mmol/L), or
  2. fasting blood glucose value ≥126 mg/dl (7 mmol/L), or
  3. a 2-hour plasma glucose ≥200 mg/dl (11.1 mmol/L) measured by Oral Glucose Tolerance Test
  Progression to diabetes will be monitored and compared between placebo and study drug treated children using the Cox regression at the 0.05 level, two-sided. With 220 children randomized over a 30 month period, and a study duration of 66 month, the study will have 86% power to detect a 50% reduction in the rate of progression to diabetes at a two-sided alpha of 0.05.
  For each secondary outcome, analyses will also be stratified by INS genotype and HLA DR4.

OTHER OUTCOMES:
Hypoglycemia | Measured at baseline (visit 1) and at subsequent change in dose (visits 2).
  Metabolic changes within two hours after receiving study drug. This will be performed at the first administration of oral insulin or placebo at each new dose (visit 1 and visit 2). At these visits, blood glucose concentrations will be measured at 0 minutes, 30 minutes, 60 minutes, and 120 minutes after receiving study drug to determine whether the treatment induces hypoglycaemia which is defined as <50 mg/dl (<2.8 mmol/L).
Adverse events | Duration of participation from study visit 1 until the end of the study (min. 36 months, max. 66 months) or drop out
  Adverse events are reported throughout the period of participation of each participant. Analysis will compare the number and frequency of adverse events during treatment with study drug (total and during each dose period) to the number and frequency of adverse events in the placebo treated children.

CONTACTS AND LOCATIONS:
Overall Officials: Anette-G. Ziegler, Prof. Dr., MD, Principal Investigator — Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München; Ezio Bonifacio, Prof. Dr., PhD, Study Chair — Paul Langerhans Institute Dresden (PLID) of the Helmholtz Zentrum München at the Universitätsklinikum Carl Gustav Carus, Technische Universität Dresden; Peter Achenbach, PD. Dr., MD, Principal Investigator — Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München; Katharina Warncke, Dr., MD, Principal Investigator — Forschergruppe Diabetes, Klinikum rechts der Isar, Techn. Universität München and Kinderklinik München Schwabing, Klinik u. Poliklinik f. Kinder- und Jugendmedizin, Klinikum Schwabing, StKM GmbH und Klinikum rechts der Isar der Techn. Universität München; Christiane Winkler, Dr., PhD, Study Chair — Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München
Locations (1):
- Forschergruppe Diabetes, Klinikum rechts der Isar, Technische Universität München, Lehrstuhl für Diabetes und Gestationsdiabetes, der Technischen Universität München, München, Deutschland (deu), Germany

REFERENCES:
- [Derived] Jacobsen LM, Schatz DA. Insulin immunotherapy for pretype 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2021 Aug 1;28(4):390-396. doi: 10.1097/MED.0000000000000648. PMID 34091488
- See also: Related Info — https://www.helmholtz-munich.de/idf